CLINICAL TRIAL: NCT03367182
Title: Real-World Effectiveness of Bevacizumab Based on AURELIA in Platinum-resistant Recurrent Ovarian Cancer
Acronym: REBECA
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2017-0748
Record Dates: First submitted 2017-11-29; First posted 2017-12-08 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Topotecan; liposomal doxorubicin; Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Weekly paclitaxel + bevacizumab
  Interventions: Drug: Weekly paclitaxel; Drug: Bevacizumab
- Topotecan + bevacizumab
  Interventions: Drug: Topotecan; Drug: Bevacizumab
- Pegylated liposomal doxorubicin + bevacizumab
  Interventions: Drug: Pegylated liposomal doxorubicin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Weekly paclitaxel — Drug: paclitaxel 80mg/m2 iv on days 1, 8, 15 and 22 of each 4-week cycle
  Groups: Weekly paclitaxel + bevacizumab
Drug: Topotecan — Drug: topotecan 4mg/m2 iv on days 1, 8 and 15 of each 4-week cycle, or 1.25 mg/kg on days 1-5 of each 3-week cycle
  Groups: Topotecan + bevacizumab
Drug: Pegylated liposomal doxorubicin — Drug: liposomal doxorubicin 40mg/m2 iv every 4 weeks
  Groups: Pegylated liposomal doxorubicin + bevacizumab
Drug: Bevacizumab — Drug: bevacizumab [Avastin] 10m/kg iv every 2 weeks or 15mg/kg iv every 3 weeks

SUMMARY:
This study will evaluate the efficacy and safety profile, response rate, progression free survival, overall survival of bevacizumab (Avastin) added to chemotherapy in patients with epithelial ovarian cancer, fallopian tube carcinoma or primary peritoneal carcinoma with disease progression within 6 months of platinum treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have histologically or cytologically confirmed recurrent epithelial ovarian cancer, fallopian tube cancer, or peritoneal cancer.
2. Patients who have platinum-resistant disease (defined as having relapsed within 6 months of her last platinum-containing regimen)
3. Patients who have underwent chemotherapy of either weekly paclitaxel + bevacizumab, topotecan + bevacizumab, pegylated liposomal doxorubicin + bevacizumab in 2nd line or 3rd line chemotherapy.

Exclusion Criteria:

1. Patients with previous treatment with bevacizumab.
2. Patients who received bevacizumab combination therapy in 4th line or more chemotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with epithelial ovarian cancer, fallopian tube carcinoma or primary peritoneal carcinoma with desease progression within 6 months of platinum treatment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 36 months
  PFS was defined as the time from the date of randomization to the first documented disease progression or death, whichever occurred first. Progression was based on tumor assessment made by the investigators according to the RECIST criteria
Incidence of Treatment-Emergent Adverse Events | 36 months
  Safety and tolerability will be assessed in deaths, laboratory data, and vital signs. Number of participants with treatment-related adverse events as assessed by CTCAE version 4.0.

SECONDARY OUTCOMES:
Response rate | 36 months
  Best Overall Confirmed Objective Response of Complete Response (CR) or Partial Response (PR) by Modified RECIST until progression reported. Objective Response was determined by the investigator using modified RECIST criteria, Version 1.0. An objective response was a complete or partial overall confirmed response as determined by investigators. CR defined as complete disappearance of all target and non-target lesions and no new lesions. PR defined as greater than or equal to (≥) 30 percent (%) decrease in the sum of appropriate diameters of all target measurable lesions, no progress in the non-measurable disease, and no new lesions.
overall survival (OS) | 36 months
  Duration of overall survival was defined as the time from randomization to death of any cause. The OS data for participants for whom no death was captured in the clinical database were censored at the last time they were known to be alive.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JY, Park JY, Park SY, Lee JW, Kim JW, Kim YB, Jeong DH, Lee KB, Kim TH, Lee IH, Choi MC, Kim KH, Kim YM, Lee YJ, Kang S; KGOG Investigators; Pujade-Lauraine E. Real-world effectiveness of bevacizumab based on AURELIA in platinum-resistant recurrent ovarian cancer (REBECA): A Korean Gynecologic Oncology Group study (KGOG 3041). Gynecol Oncol. 2019 Jan;152(1):61-67. doi: 10.1016/j.ygyno.2018.10.031. Epub 2018 Nov 6. PMID 30409490